CLINICAL TRIAL: NCT04864964
Title: The Value of Sensory Index in Predicting the Success of Radiofrequency Treatment of Trigeminal Neuralgia: A Retrospective Study
Brief Title: the Value of Sensory Index in Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Associate Professor of Anesthesia, intensive care and Pain releif, National Cancer Institute, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ehab-Hossam trigeminal
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined conventional and pulsed radiofrequency of trigeminal nerve nucleus (Other): The technique of the CCPRF is described as follows;
  1. the classic Hartle technique is used to reach the Gasserian ganglion
  2. Sensory stimulation with the RF equipment is conducted and parathesia of the affected branch is achieved at 0.1-0.2 V (50 Hz), keeping in mind that the mandibular part of the Gasserian ganglion is ventrolateral and the ophthalmic rootlets are postrolateral. Motor pre-stimulation (2 Hz) is achieved with masseter contraction at 0.1-0.3 V .
  3. After sensory and motor stimulation, RF therapy is conducted by use of the RF generator , in the sequence:
     * Conventional RF 1st lesion at 60 °C for 60 s then 2nd lesion at 65°C for 60 seconds then 3rd lesion at 70°C for 60 seconds
     * Finally, PRF is applied for 360 second repeated at 45 V, with a pulse width of 10 ms and a pulse frequency of 4 Hz. The cut-off needle tip temperature is set at 42 °C.
  4. Before withdrawal of needle 1 cc xylocaine 1% + 0.5 cc dexamethasone 4mg to be given .
  Interventions: Procedure: combined conventional and pulsed radiofrequency (CCPRF)

INTERVENTIONS:
Procedure: combined conventional and pulsed radiofrequency (CCPRF) — Patients with trigeminal neuralgia who underwent combined conventional and pulsed radiofrequency (CCPRF) for treatment of pain.

SUMMARY:
Interventional therapies for Trigeminal Neuralgia are of variable efficacy and safety, and have different results for different periods of time before the recurrence of symptoms. Interventional therapy for TN is either destructive with trigeminal nerve sensory function destroyed intentionally or non-destructive with decompression of the trigeminal nerve and preservation of its regular function. The most common procedures in treating TN pain are the use of radiofrequency (RF). the aim of this study is to assess the possible value of motor index as a prediction of success of radiofrequency lesioning of the Gasserian ganglion during treatment of trigeminal neuralgia.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is defined by the International Headache Society (IHS) as "unilateral disorder characterized by brief electric shock-like pains, abrupt in onset and termination, and limited to the distribution of one or more divisions of the trigeminal nerve". It is considered the worst type of facial pain and described as intense, sharp, stabbing, and shooting like electric shock pain. It can be triggered by touch, chewing, laughing, shaving or face wash .

The IHS suggests a classification of TN as either classic (essential or idiopathic) TN (CTN) or symptomatic TN (STN; pain indistinguishable from that of CTN, but caused by a demonstrable structural lesion other than vascular compression).Treatment of TN is conservative, surgical or interventional. Pharmacotherapy with carbamazepine is tried early in cases of TN but has many side effects .Other medications can be used in the treatment of TN, include oxycarbazepine, gabapentin, pregabalin, baclofen, valproate, clonazepam, phenytoin, and lamotrigime .

The most clinically appropriate treatment includes surgical microvascular decompression (MVD), stereotactic radiation therapy, gamma knife (SGK), percutaneous balloon decompression, percutaneous glycerol rhizolysis, percutaneous radiofrequency (RF) of the Gasserian ganglion (GG), and GG stimulation and neuromodulation. Interventional therapies for TN are of variable efficacy and safety, and have different results for different periods of time before the recurrence of symptoms. Interventional therapy for TN is either destructive with trigeminal nerve sensory function destroyed intentionally or non-destructive with decompression of the trigeminalnerve and preservation of its regular function. The most common procedures in treating TN pain are the use of radiofrequency (RF) .

Radiofrequency thermos-coagulation of the GG is thought to selectively destroy the pain fibers by thermos-coagulation at > 65°C , that helps reduce pain and prevent triggering, but can cause bothersome dysesthesia. Another method, pulsed radiofrequency (PRF) which defined as the delivery of short pulses of RF via a needle tip, thereby a short exposure at the same temperature will result in less thermal tissue destruction (6).

Combined conventional and pulsed radiofrequency (CCPRF) achieved comparable pain relief to PRF treatment alone in patients with chronic pain, the combination of PRF and CRF would increase the effect of CRF and reduce the need for long-duration CRF (LCRF) and its attendant side effects .

The main objective of this study is to assess the possible value of motor index as a prediction of success of radiofrequency lesioning of the Gasserian ganglion during treatment of trigeminal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trigeminal neuralgia, diagnosed in accordance with the International Headache Society (7) and with a visual analogue score (VAS) for pain of at least 7 or more for a minimum of 3 months before the intervention .
* Patients on a stable analgesic regimen for 2 weeks (consisting of at least two analgesics, including anticonvulsants) before the intervention .
* Patients examined by use of MRI/A of the brain to exclude secondary neuralgia.

Exclusion Criteria:

* Patients with severe mental or psychiatric disorders
* Patients with history of drug abuse, high intracranial tension and history of MVD, SGK, balloon compression, RF treatment, or glycerol injection
* The possibility of vascular loop compression and other causes of TN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Motor index | 2 weeks
  Change of the visual analogue scale score, from 0 to 100 , where 100 means worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
contacts personal details are not planned to be shared but the results can be shared after publication

REFERENCES:
- See also: efficacy of Pulsed Radiofrequency Stimulation in Patients with Peripheral Neuropathic Pain: A Narrative Review — http://painphysicianjournal.com/current/pdf?article=NTIxNQ%3D%3D&journal=111